CLINICAL TRIAL: NCT06138808
Title: Prognostic Value of the 5-SENSE Score to Predict Focality of the Seizure-onset Zone as Assessed by Stereo-electroencephalography - a Prospective Multicenter Validation Study
Brief Title: 5-SENSE Score Validation Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Christian Doppler University Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00113692
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy Intractable
Keywords: epilepsy; surgery; stereo-electroencephalography
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stereoelectroencephalography (SEEG): Participants undergoing SEEG as part of standard of care.
  Interventions: Other: Stereoelectroencephalography (SEEG)
- Control Group: Participants not undergoing SEEG as part of standard of care.

INTERVENTIONS:
Other: Stereoelectroencephalography (SEEG) — Participants will under Stereoelectroencephalography (SEEG) as part of standard of care. This is not assigned by the protocol.
  Groups: Stereoelectroencephalography (SEEG)

SUMMARY:
The purpose of this study is to assess how well a new scoring system called the 5-SENSE score can predict where seizures start in the brain using Stereoelectroencephalography (SEEG). The 5-SENSE Score is a 5-point score based on routine presurgical work-up, designed to assist in predicting whether SEEG can identify a focal seizure onset zone, thereby sparing patients the risk of undergoing this invasive diagnostic procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 15 years or older in whom no direct surgical approach can be offered and who are discussed in the multidisciplinary team discussion
* availability of complete non-invasive presurgical work-up (including high-resolution MRI according to the in-center epilepsy protocol, video-telemetry with the recording of a minimum of one habitual clinic and EEG seizure, available as original files for review)

Exclusion Criteria:

* no telemetry/scalp EEG in center
* no protocol MRI in center
* subdural/GRID electrodes

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients will be prospectively recruited at 20-25 epilepsy centers from North America, Europe, Australia and Asia.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Specificity of the 5-SENSE score for the identification of a focal SOZ on SEEG | At time of SEEG, up to approximately 1 month
  Prospective validation of the predictive value of the 5-SENSE score to identify a focal seizure onset zone (SOZ) in an independent patient sample. Measured for participants undergoing SEEG.
Sensitivity of the 5-SENSE score for the identification of a focal SOZ on SEEG | At time of SEEG, up to approximately 1 month
  Prospective validation of the predictive value of the 5-SENSE score to identify a focal seizure onset zone (SOZ) in an independent patient sample. Measured for participants undergoing SEEG.
Positive predictive value of the 5-SENSE score for the identification of a focal SOZ on SEEG | At time of SEEG, up to approximately 1 month
  Measured for participants undergoing SEEG
Negative predictive value of the 5-SENSE score for the identification of a focal SOZ on SEEG | At time of SEEG, up to approximately 1 month
  Measured for participants undergoing SEEG

SECONDARY OUTCOMES:
Specificity of the 5-SENSE score augmented by information from auxiliary diagnostic methods for the identification of a focal SOZ on SEEG | At time of SEEG, up to approximately 1 month
  For participants undergoing SEEG, information from auxiliary diagnostic methods, performed routinely during presurgical evaluation, namely FDG-PET, electrical source imaging (ESI) and/or magnetic source imaging (MSI) and ictal HMPAO-SPECT will be analyzed. The investigators will assess whether addition of those variables to the 5-SENSE Score could enhance score performance with higher specificity for identifying a focal SOZ
Sensitivity of the 5-SENSE score augmented by information from auxiliary diagnostic methods for the identification of a focal SOZ on SEEG | At time of SEEG, up to approximately 1 month
  For participants undergoing SEEG, information from auxiliary diagnostic methods, performed routinely during presurgical evaluation, namely FDG-PET, electrical source imaging (ESI) and/or magnetic source imaging (MSI) and ictal HMPAO-SPECT will be analyzed. The investigators will assess whether addition of those variables to the 5-SENSE Score could enhance score performance with higher sensitivity for identifying a focal SOZ
Concordance of the 5-SENSE Score with the decision whether to proceed with SEEG or not | At enrollment
  Before SEEG, the decision whether to proceed with SEEG or not is made blinded from the 5- SENSE Score in a Multidisciplinary Team Discussion (MTD). Following the decision, the 5-SENSE Score will be calculated for each participant by the principal investigator. Concordance of the 5-SENSE Score with the decision made in the MTD will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Frauscher, MD PD, Principal Investigator — Duke University; Alexandra Astner-Rohracher, Principal Investigator — Christian Doppler University Hospital Paracelsus Medical University Salzburg and Centre for Cognitive Neuroscience Salzburg
Locations (19):
- United States (4):
  - University of Florida College of Medicine, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Duke University Health System, Durham, North Carolina
  - Presbyterian-Shadyside Hospital, Pittsburgh, Pennsylvania
- Australia (3):
  - Monash University, Melbourne, Victoria
  - Mater Health, Brisbane
  - Alfred Health, Melbourne
- Christian Doppler University Hospital Paracelsus Medical University Salzburg and Centre for Cognitive Neuroscience Salzburg, Salzburg, Austria
- Canada (2):
  - Dalhousie Universiry and Hospital, Dalhousie, Nova Scotia
  - Wester University, London, Ontario
- Departmet of Neurology, Masaryk University Brno, Brno, Czechia
- Danish Epilepsy Centre, Aarhus Universitets Hospital, Aarhus, Denmark
- France (2):
  - Grenoble Institute of Neurosciences, Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Epilepsy Department University Hospitals of Marseille, Marseille
- Epilepsy Centre, University Hospital Freiburg, Freiburg im Breisgau, Germany
- University School of Medicine Kyoto, Kyoto, Japan
- "Carol Davila" University of Medicine and Pharmacy, Bucharest, Romania
- Hospital Universitario y Politecnico La Fe, Valencia, Spain
- Department of Clinical Neurosciences chez CHUV; Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Astner-Rohracher A, Ho A, Archer J, Bartolomei F, Brazdil M, Cacic Hribljan M, Castellano J, Dolezalova I, Fabricius ME, Garces-Sanchez M, Hammam K, Ikeda A, Ikeda K, Kahane P, Kalamangalam G, Kalss G, Khweileh M, Kobayashi K, Kwan P, Laing JA, Leitinger M, Lhatoo S, Makhalova J, McGonigal A, Mindruta I, Mizera MM, Neal A, Oane I, Parikh P, Perucca P, Pizzo F, Rocamora R, Ryvlin P, San Antonio Arce V, Schuele S, Schulze-Bonhage A, Suller Marti A, Urban A, Villanueva V, Vilella Bertran L, Whatley B, Beniczky S, Trinka E, Zimmermann G, Frauscher B. Prognostic value of the 5-SENSE Score to predict focality of the seizure-onset zone as assessed by stereoelectroencephalography: a prospective international multicentre validation study. BMJ Neurol Open. 2024 Aug 21;6(2):e000765. doi: 10.1136/bmjno-2024-000765. eCollection 2024. PMID 39175939